CLINICAL TRIAL: NCT04337138
Title: Characteristics, Treatment Patterns, and Clinical Outcomes in Acute Myeloid Leukemia (AML) Patients Using Mylotarg - a US Real-World Study Using Electronic Medical Record Data
Brief Title: A Study Of Treatment Patterns And Clinical Outcomes In Patients Diagnosed With Acute Myeloid Leukemia Who Received Mylotarg in the Real-World
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1761033
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AML; Mylotarg; gemtuzumab
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Gemtuzumab Ozogamicin — Gemtuzumab Ozogamicin (Mylotarg) administered in any form or combination
  Other Names: Mylotarg

SUMMARY:
The aim of this observational study is to describe treatment patterns and effectiveness outcomes in a sample of oncology patients treated for AML with Mylotarg through up to two additional relapsed/refractory (R/R)-based lines of therapy (through third-line therapy). The study will use United States oncology electronic medical record (EMR) data. All study data are secondary data and will have been collected retrospectively from existing clinical data originally collected as part of routine care.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of acute myeloid leukemia (AML) on or after 01 December 2014 through Clinical Research Nurse (CRN) review of provider documentation of AML diagnosis in the medical record;
* Receipt of Mylotarg at any point during first three lines of therapy following initial AML diagnosis;
* Age greater than or equal to 18 years at initial diagnosis of AML.

Exclusion Criteria:

- Record of 1 or more of the following confounding diagnoses at any point before or after AML diagnosis: Acute lymphoblastic leukemia; acute promyelocytic leukemia, aggressive systemic mastocytosis; hypereosinophilic syndrome and/or chronic eosinophilic leukemia; dermatofibrosarcoma protuberans; gastrointestinal stromal tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients diagnosed with AML who, at any point on or after September 1, 2017 received Mylotarg, alone or in combination with other agents for newly diagnosed or relapsed refractory AML.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2020-04-07 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1761033

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, data for participants was collected retrospectively through the United States oncology electronic medical record data available to Concerto HealthAI, including data from CancerLinQ-affiliated practices (referred as definitive oncology dataset).
Groups:
- Mylotarg: Participants with confirmed diagnosis of Acute Myeloid Leukemia (AML) on or after 01 December 2014, who received Mylotarg (Gemtuzumab ozogamicin [mean number of doses of gemtuzumab administered = 1 per participant]) from 2017 to 2020 in real-world clinical setting (i.e. treated in clinical practice and in a non-trial setting) were included in this retrospective study and their data from definitive oncology dataset was retrospectively assessed in this study of up to 4 months.
Period: Overall Study
Arm/Group | Mylotarg
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants who were included in this study.
Arm/Group | Mylotarg
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.9 (14.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 26
  More than one race | 0
  Unknown or Not Reported | 4
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kilogram/meters^2] | 29.7 (5.88)
Insurance Status [Count of Participants; unit: Participants] — Here, number of participants with their insurance status as 'private only, public only, both (public and private insurance), neither (unknown or undocumented)' were reported. Private only insurance was purchased by the participants. Public only insurance was provided by the federal or state funds.
  Participants
    Private Insurance, No Public Insurance | 4
    Public Insurance, No Private Insurance | 1
    Public and Private Insurance | 5
    Unknown/Undocumented | 22
Height of Participants [Mean (Standard Deviation); unit: Inches] — Population: Here 'number analyzed" signifies participants evaluable for this baseline measure.
  Inches
    number analyzed (Participants) | 30
    (all) | 67.5 (3.73)
Body Weight [Mean (Standard Deviation); unit: Pounds] | 185.1 (52.71)
Region of Residence [Count of Participants; unit: Participants] — Here, number of participants were classified in 5 categories (Midwest, northeast, south, west and undocumented [unknown] region) according to their region of residence.
  Participants
    Midwest | 5
    Northeast | 1
    South | 4
    West | 2
    Undocumented Region | 20
Number of Participants With Comorbidities [Count of Participants; unit: Participants] — Here, number of participants were classified in 4 categories (congestive heart failure, connective tissue disease, diabetes and myocardial infarction) according to different type of comorbid condition. Population: Here "number analyzed" signifies participants evaluable for this baseline measure.
  Participants
    number analyzed (Participants) | 15
    Congestive Heart Failure | 1
    Connective Tissue Disease | 2
    Diabetes | 11
    Myocardial Infarction | 1
Mean Charlson Comorbidity Index of Participants [Mean (Standard Deviation); unit: Units on a scale] — Charlson Comorbidity Index scored the cumulative severity of a participant's comorbidities. Total score ranged from 0 to 9. A score of zero indicated that no comorbidities were found. The higher the score, the more likely the cumulative severity of a participant's comorbidities. Population: Here "number analyzed" signifies participants evaluable for this baseline measure.
  Units on a scale
    number analyzed (Participants) | 14
    (all) | 1.1 (0.27)
Number of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — ECOG PS was used to assess physical health of participant, ranged from 0 (most active) to 5 (dead) where 0=fully active, able to carry on all pre-disease performance without restriction; 1=restricted in physically strenuous activity, ambulatory, able to carry out light or sedentary work; 2=ambulatory, capable of all self-care, unable to carry out any work activity, up greater than (>)50 percent (%) of waking hours; 3=capable of only limited self-care, confined to bed or chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed or chair; 5=dead.
  Participants
    0 | 4
    1 | 5
    2 | 3
    3 | 1
    4 | 0
    5 | 0
    Undocumented ECOG | 19
AML Stage at Index Date [Count of Participants; unit: Participants] — Here, number of participants were classified according to their AML type. Index date was defined as the date of initial AML diagnosis.
  Participants
    De Novo | 22
    Secondary | 8
    Undocumented | 2
Number of Participants With Results for Cytogenetic/FISH Testing at Initial AML Diagnosis [Count of Participants; unit: Participants] — Here, number of participants were classified according to positive results (if they had test result data available and denoted as "yes") and and negative results (if they did not had test result data and denoted as "no") in cytogenetic/ Fluorescence in situ Hybridization (FISH) testing. Cytogenetic/FISH testing included: t(6;9)(p23:q34.1), t(v;11q23.3), t(9;22)(q34.1;q11.2), inv(3)(q21.3q26.2) or t(3;3)(q21.3;q26.2), -5 or del(5q); -7; -17/abn(17p), complex karyotype, monosomal karyotype, t(8;21)(q22;q22.1), inv(16)(p13.1q22) and t(16;16)(p13.1;q22) tests.
  Participants
    t(6;9)(p23:q34.1) Testing: Yes | 0
    t(6;9)(p23:q34.1) Testing: No | 32
    t(v;11q23.3) Testing: Yes | 0
    t(v;11q23.3) Testing: No | 32
    t(9;22)(q34.1;q11.2) Testing: Yes | 0
    t(9;22)(q34.1;q11.2) Testing: No | 32
    inv(3)(q21.3q26.2)³ or t(3;3)(q21.3;q26.2) Testing: Yes | 2
    inv(3)(q21.3q26.2)³ or t(3;3)(q21.3;q26.2) Testing: No | 30
    -5 or del(5q); -7; -17/abn(17p) Testing: Yes | 1
    -5 or del(5q); -7; -17/abn(17p) Testing: No | 31
    Complex karyotype Testing: Yes | 1
    Complex karyotype Testing: No | 31
    Monosomal karyotype Testing: Yes | 1
    Monosomal karyotype Testing: No | 31
    t(8;21)(q22;q22.1) Testing: Yes | 3
    t(8;21)(q22;q22.1) Testing: No | 29
    inv(16)(p13.1q22)¹ or t(16;16)(p13.1;q22) Testing: Yes | 3
    inv(16)(p13.1q22)¹ or t(16;16)(p13.1;q22) Testing: No | 29

OUTCOME MEASURES:

1. Primary Outcome: Real-World Event-Free Survival (rwEFS)
Description: rwEFS defined as time from treatment initiation date (for first line of Mylotarg-containing therapy) to date of treatment failure (TF), relapse from complete response (CR) or better, death from any cause, whichever came first. TF defined as failure to achieve CR or better following up to 3 cycles of Mylotarg. Time origin for rwEFS was start of Mylotarg in first line of therapy in which it was used. Terminal event for analysis of rwEFS was earlier of treatment failure, relapse from CR or better, death. CR is defined as having less than (<) 5% blasts in the bone marrow and 0% blasts in the peripheral blood. Real-world setting signifies participants treated in clinical practice and in a non-trial setting.
Time Frame: From treatment initiation date to date of TF, relapse from CR or better, death from any cause, whichever came first (maximum duration of 3 years)
Population: Analysis population included all participants included in this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mylotarg
Number analyzed (Participants) | 32
months | 1.66 [0.9 to 4.8]

2. Primary Outcome: Real-World Relapse Free Survival (rwRFS)
Description: rwRFS was defined as the time from the treatment initiation date (during the first line of Mylotarg-containing therapy) to the date of a relapse event, or death from any cause, whichever came first. The time origin for rwRFS was the start of Mylotarg in the first line of therapy in which it was used. Real-world setting signifies participants treated in clinical practice and in a non-trial setting.
Time Frame: From the treatment initiation date (during the first line of Mylotarg-containing therapy) to the date of a relapse event, or death from any cause, whichever came first (maximum duration of 3 years)
Population: Analysis population included all participants included in this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mylotarg
Number analyzed (Participants) | 32
months | 4.87 [2.6 to 8.2]

3. Primary Outcome: Real-World Overall Survival (rwOS)
Description: rwOS was defined as the time from the start of the first Mylotarg use till the date of death. Participants who were not indicated to be deceased in clinical records or Social Security Disability Insurance (SSDI) records were censored for rwOS analysis as of the later of 1) the latest date known alive within the clinical record, 2) 4 months prior to the date of most recent SSDI update. Real-world setting signifies participants treated in clinical practice and in a non-trial setting.
Time Frame: From the start of the first Mylotarg use till death (maximum duration of 3 years)
Population: Analysis population included all participants included in this study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mylotarg
Number analyzed (Participants) | 32
months | 6.15 [3.1 to NA] — The upper limit of 95% confidence interval was not estimable due to small sample size as a result of censoring.

4. Primary Outcome: Number of Participants With First Positive Response
Description: First positive response was assessed by physician as first response from any of the following: CR, partial response (PR), stable disease (SD) and progressive disease (PD). CR is defined as having < 5% blasts in the bone marrow and 0% blasts in the peripheral blood. PR is defined as having 5 to 25% bone marrow blasts with > 50% reduction in blasts and peripheral blood count recovery. SD is defined as having no change in bone marrow blasts. PD is defined as having relapse following response. Participant for whom record did not indicate one of these classification classed as not evaluable (NE).
Time Frame: From the first qualifying Mylotarg-containing line of therapy to the end of the third line of therapy or the end of record, whichever occurs first (maximum duration of 3 years)
Population: Analysis population included all participants included in this study. Here, 'number analyzed' signifies participants evaluable for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Mylotarg
Number analyzed (Participants) | 32
Participants
  First line (1L) Therapy: number analyzed (Participants) | 16
  First line (1L) Therapy: CR | 9
  First line (1L) Therapy: NA-Participant had SD, PD, NE, no documentation of response assessment or other negative response | 7
  First line (1L) Therapy: PR | 0
  Second line (2L) Therapy: number analyzed (Participants) | 8
  Second line (2L) Therapy: CR | 2
  Second line (2L) Therapy: NA-Participant had SD, PD, NE, no documentation of response assessment or other negative response | 5
  Second line (2L) Therapy: PR | 1
  Third line (3L) Therapy: number analyzed (Participants) | 8
  Third line (3L) Therapy: CR | 0
  Third line (3L) Therapy: NA-Participant had SD, PD, NE, no documentation of response assessment or other negative response | 5
  Third line (3L) Therapy: PR | 3

5. Other Pre Specified Outcome: Duration of Therapy
Description: Duration of therapy was time from the initiation of Mylotarg to the last date of Mylotarg therapy, regardless of line of therapy (duration could continue into subsequent lines of therapy), study end date, or death, whichever came first.
Time Frame: From the initiation of Mylotarg to the last date of Mylotarg therapy (maximum duration of 3 years)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Mylotarg
Number analyzed (Participants) | 32
months
  Mylotarg in 1L therapy: number analyzed (Participants) | 16
  Mylotarg in 1L therapy | 1.6 (2.13)
  Mylotarg in 2L therapy: number analyzed (Participants) | 8
  Mylotarg in 2L therapy | 1.2 (1.36)
  Mylotarg in 3L therapy: number analyzed (Participants) | 8
  Mylotarg in 3L therapy | 1.0 (1.99)

6. Post Hoc Outcome: rwEFS in De-Novo AML Participants Using a Closer-to-Typical Combination of Mylotarg + Chemotherapy as 1L Therapy
Description: rwEFS defined as time from treatment initiation date (for first line of Mylotarg-containing therapy) to date of TF, relapse from CR or better, death from any cause, whichever came first. TF defined as failure to achieve CR or better following up to 3 cycles of Mylotarg. Time origin for rwEFS was start of Mylotarg in first line of therapy in which it was used. Terminal event for analysis of rwEFS was earlier of treatment failure, relapse from CR or better, death. CR is defined as having < 5% blasts in the bone marrow and 0% blasts in the peripheral blood. Real-world setting signifies participants treated in clinical practice and in a non-trial setting.
Time Frame: as for outcome 1
Population: Analysis population included all participants included in this study. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Mylotarg
Number analyzed (Participants) | 7
months | 6.15 [0.5 to NA] — 95% confidence interval upper limit was not estimable due to very less number of participants.

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events not collected during the study
Description: This study involved data that existed as structured data by the time of study start. In these data sources, individual participant data were not retrieved or validated, and it was not possible to link a particular product and medical event for any individual. Thus, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) was not met, hence, safety data was not planned to be collected and reported.
Arm/Group | Mylotarg
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT04337138/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/38/NCT04337138/SAP_001.pdf